CLINICAL TRIAL: NCT03791359
Title: Warangal Area Out of Hospital Cardiac Arrest Registry-A Pilot Project In India (WACAR)
Brief Title: A Pilot Project of Out Of Hospital Cardiac Arrests in Warangal Area,Telangana,India
Acronym: WACAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SRINIVAS RAMAKA (Other)
Responsible Party: Sponsor-Investigator, SRINIVAS RAMAKA, Principal Investigator, Srinivasa Heart Centre
Organization: Srinivasa Heart Centre (Other)
Other Study IDs: KIEC/KMC/NCT/NIS/2018/CAR01
Record Dates: First submitted 2018-12-31; First posted 2019-01-02 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Out- of- Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CardioPulmonary Resuscitation — Whether the victim received CPR as per standard protocol.

SUMMARY:
This Pilot project is an observational study of a cohort of participants (victims) of Out of Hospital Cardiac Arrests in Warangal area ,Telangana ,India .

Started on January 1,2018 to December 2018.

DETAILED DESCRIPTION:
Introduction and Background:Cardiac arrest is an important public health problem worldwide.Registries on Out Of Hospital Cardiac arrest(OOHCA) not only contribute to research and surveillance but also provide inputs to improve the links in the Chain of Survival.Whereas various registries on OOHCA exist and are ongoing globally ,registries and studies on OOHCA are limited in India.The awareness on Cardiovascular Health, Cardiac Arrest and CPR is less in India when compared to some developed countries.A study done earlier noted the lack of awareness on Cardiovascular Health,cardiac arrest and CPR in a cohort of Indian population.This study pointed the need to increase awareness on CV health,cardiac arrest and CPR among Indian population(abstract presented by Dr Srinivas Ramaka at the World Congress of Cardiology,2016).There is a dire need to improve the survival of victims of OOHCA in India.

With this background and understanding,the need for a Registry on OOHCA ,the Warangal Area Out Of Hospital Cardiac Arrest Registry has been initiated in January 2018 as a Pilot study in India.

Objectives:1.To collect available OOHCA data for one year from a selected geographical area in India following an International standard format(Utstein Template) tailored to India.

2.To compile reports which might be useful to improve the links in the survival of OOHCA victims.

Methods and study design:This is an Observational study of a cohort of Out of Hospital cardiac arrest victims. Geographical area:Warangal and surroundings ,Telangana state. Time frame--January 1 ,2018 to December 31,2018.As it is both a surveillance and research study,the project is proposed to be continued mostly for another year 2019 depending on logistic support and feasibility.

Sources of data:Mahatma Gandhi Memorial Hospital,participating local hospitals and practising physicians,reports from local media,local governmental agencies,births and deaths department of local Municipal Corporation and district medical and health officials.MGM Hospital is a secondary care govt hospital catering to the medical needs of Warangal and surrounding districts.Data of victims brought in cardiac arrest or declared dead on arrival is collected from the Casualty or Emergency dept .Missing data or additional information is collected telephonically from the victim's relatives and attendants.The local legal and ethical guidelines are followed in collecting the data.Data is collected on a standard report form /Online fillable pdf which includes the variables as mentioned in the data collection form,participants/cohorts of victims of OOHCA,definition of OOHCA,inclusion criteria,sources of information collected in person or telephonically,consent,methods of selection of participants and methods of followup.Data is entered in standard excel format and will be analyzed according to appropriate/standard statistical methods.Permission from the hospital administration and all concerned is taken prior.At present there is no funding for the project.Dr Srinivas Ramaka is the Principal Investigator. Dr Vemuri S Murthy from USA is the coinvestigator in this project.

Acknowledgements:Superintendent,MGM Hospital,Warangal,DMHO ,Warangal,Registrar ,Births and Deaths,Warangal,doctors and Staff,Casualty,MGM Hospital,.Dept of Medicine,MGM Hospital,local medical and pharmacy students, local media, and relatives and attendants of victims of OOHCA.

ELIGIBILITY:
Inclusion Criteria:

* All participants(victims) of Out Of Hospital Cardiac Arrest above 18 years.

Exclusion Criteria:

*Participants(victims) of OOHCA whose data is not available or whose attendants are unwilling to share the data are excluded from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of victims of Out of Hospital Cardiac arrests which occur in Warangal Area,Telangana State ,India from January 1 2018 to December 2018.Survival outcomes and other variables as mentioned in the study protocol are studied.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Survival with good neurological state of OOHCA victims | From cardiac arrest upto 3 months and beyond.
  Percentage of those who survived an instance of OOHCA with good neurological outcome

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Ramaka, MD, Principal Investigator — Srinivasa Heart Centre; Vemuri S Murthy, MD, Study Chair — University of Illinois, Chicago,Illinois
Locations (1):
- Srinivasa Heart Centre, Warangal, Telangana, India

IPD SHARING:
Plan to Share IPD: Undecided
Will inform later as this is a Pilot Study in India.